CLINICAL TRIAL: NCT05818982
Title: A Multicenter, Open-label, Randomized, Controlled Phase II Study to Evaluate the Efficacy and Safety of Afatinib Versus Irinotecan as a Second-line and Above Treatment for Advanced ALTRK-negative ESCC
Brief Title: To Evaluate the Efficacy and Safety of Afatinib for Advanced ALTRK-negative ESCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESCC-ALTRK
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Advanced Esophageal Squamous Cell Carcinoma
MeSH Terms: interventions — Afatinib; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): Group A received afatinib (40 mg oral/day) every 6 weeks
  Interventions: Drug: Afatinib
- Cohort B (Active Comparator): Group B received irinotecan (140-180mg/m2 intravenous) every 2 weeks
  Interventions: Drug: Irinotecan

INTERVENTIONS:
Drug: Afatinib — Afatinib will be administered orally at 40 mg per day (qd) in each 6-week cycle.
  Arms: Cohort A
Drug: Irinotecan — Irinotecan, intravenous drip, 140-180mg/㎡, D1, Q14D
  Arms: Cohort B

SUMMARY:
This is a phase II study to evaluate the effectiveness and safety of Afininib compared to irinotecan in the 3-gene RNA sequencing (ALTRK) negative advanced esophageal squamous squamous carcinoma.

DETAILED DESCRIPTION:
Participants were assigned to either group A or group B at 2:1 randomization (block randomization). Group A received afatinib (40 mg orally/day) every 6 weeks; Group B received irinotecan (140-180mg/m2 intravenous) every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to participate and sign the informed consent form in writing;
2. Age: 18-75 years old;
3. No gender limit;
4. Esophageal squamous cell carcinoma diagnosed by pathology;
5. The results of 3-gene RNA sequencing (ALTRK) in tumor tissue were negative;
6. Imagingly confirmed unresectable advanced esophageal squamous cell carcinoma;
7. Failure of previous platinum-containing regimens and immunotherapy regimens (PD-1/PD-L1 monoclonal antibody);
8. At least one measurable lesion (according to RECIST1.1 criteria) or non-measurable lesion that can be evaluated, with imaging diagnosis ≤ 21 days from enrollment;
9. Estimated survival≥ 3 months;
10. General Physical Condition (ECOG) 0-1;
11. Sufficient bone marrow hematopoietic function (within 7 days): hemoglobin ≥ 9 g/dL, white blood cell ≥ 3.0×10^9/L, neutrophil ≥1.5×10^9/L, platelet ≥ 100×10^9/L; Normal liver and kidney function (within 14 days): TBIL ≤ 1.5 times the upper limit of normal; ALT and AST ≤ 2.5 times the upper limit of normal, and if liver metastases are present, ≤ 5 times the upper limit of normal; Creatinine ≤ 1.5 times the upper limit of normal;

Exclusion Criteria:

1. Those who are currently receiving other effective programs;
2. Patients who have participated in other clinical trials within 4 weeks before enrollment;
3. There is no measurable tumor foci, such as fluid accumulation in the body cavity or diffuse infiltration of organs;
4. Those who have received radiotherapy for measurable lesions;
5. Previous anti-EGFR monoclonal antibody or EGFR-TKI treatment;
6. Patients with other primary malignant tumors other than esophageal cancer at the same time, except for cured skin basal cell carcinoma and cervical carcinoma in situ;
7. Clinically significant cardiovascular diseases, such as heart failure (NYHA GRADE III-IV), uncontrolled coronary heart disease, cardiomyopathy, arrhythmia, uncontrolled hypertension or history of myocardial infarction within the past 1 year;
8. Neurological or psychiatric abnormalities affecting cognitive ability, including central nervous system metastases;
9. Active severe clinical infection (grade >2 NCI-CTCAE version 5.0) within 14 days prior to enrollment, including active TB;
10. Known or reported HIV infection or active hepatitis B or C;
11. Uncontrolled systemic diseases, such as poorly controlled diabetes;
12. History of interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or evidence of interstitial lung disease on baseline chest x-ray/CT;
13. Keratitis, ulcerative keratitis or severe dry eye;
14. Known hypersensitivity or anaphylaxis to any component of the investigational drug;
15. Pregnancy (determined by serum β-chorionic gonadotropin test) or breastfeeding;
16. The investigator determines that there are abnormal heart or lung or kidney or liver function that is not suitable for the treatment of this study;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-02-09 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  PFS is defined as the time from the first dose to the date of the disease progression or death from any cause.

SECONDARY OUTCOMES:
Objective response rate | 2 years
  The Objective Response Rate (ORR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.
Disease control rate | 2 years
  Disease control rate (DCR) is the percentage of participants who achieved Complete Response (CR) or Partial Response (PR) or Stable disease (SD) based on RECIST version 1.1.
Overall survival | 2 years
  OS is defined as the time from the first dose to the date of death due to any cause.
Adverse Events | 2 years
  Incidence and severity of adverse events.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, China, Beijing
  - First Hospital of Xiamen University Affiliated Hospital,Xiamen,China, Xiamen
  - Xinxiang Central Hospital of Henan Province, Xinxiang, China, Xinxiang

IPD SHARING:
Plan to Share IPD: No